CLINICAL TRIAL: NCT01278069
Title: PET-AML - Value of 18FDG-PET-CT in Patients With AML for Detection of Extramedullary AML Manifestations
Brief Title: PET-CT in AML for Detection of Extramedullary AML Manifestations
Acronym: PETAML
Status: Completed | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Principal Investigator, Friedrich Stölzel, M.D., PET-AML - Value of 18FDG-PET-CT in Patients With AML for Detection of Extramedullary AML Manifestations, Technische Universität Dresden
Other Study IDs: TUD-PETAML-043
Record Dates: First submitted 2011-01-14; First posted 2011-01-17 (Estimated); Last update posted 2013-09-18 (Estimated); Status verified 2013-09

CONDITIONS: Newly Diagnosed or Relapsed Acute Myeloid Leukemia
Keywords: Acute myeloid Leukemia; Myeloid Sarcoma; Extramedullary Acute myeloid Leukemia; 18FDG-PET-CT
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Sarcoma, Myeloid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Myeloid Sarcoma (or granulocytic Sarcoma or Chloroma) is well defined by the WHO. However, there are currently no data about the prevalence, sites of occurence and thr prognostic value for patients with AML with this finding. Information about this condition is based on retrospective analyses since there have been no studies trying to define the role of myeloid sarcoma in AML so far. This observational trial will include adult patients with newly diagnosed and relapsed AML in order to perform 18FDG-PET-CT imaging prior to induction chemotherapy. Furthermore, a second 18FDG-PET-CT will be performed after induction chemotherapy to define the responsiveness of these tumors to chemotherapy. The primary endpoint of this study is the prevalence of 18FDG-PET-CT positive extramedullary AML manifestations (myeloid sarcoma) in patients with newly diagnosed or relapsed AML.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed or relapsed AML
* AML FAB M0-2, M4-7
* Signed informed consent after patient information
* Male and female patients with AML age 18-80
* 18FDG-PET-CT is available within a period of 5 days after diagnosis of AML

Exclusion Criteria:

* AML FAB M3 (Promyelocytic Leukemia)
* lacking willingness to cooperate
* pregnancy or insufficient contraception
* 18FDG-PET-CT is not available within a period of 5 days after diagnosis of AML
* Medical condition of the patients requires an immediated start of chemotherapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients or Outpatients with newly diagnosed or relapsed AML AML
Sampling Method: Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2011-02; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medizinische Klinik und Poliklinik I, Universitätsklinikum Carl Gustav Carus, Dresden, Saxony, Germany

REFERENCES:
- [Derived] Stolzel F, Rollig C, Radke J, Mohr B, Platzbecker U, Bornhauser M, Paulus T, Ehninger G, Zophel K, Schaich M. (1)(8)F-FDG-PET/CT for detection of extramedullary acute myeloid leukemia. Haematologica. 2011 Oct;96(10):1552-6. doi: 10.3324/haematol.2011.045047. Epub 2011 Jun 17. PMID 21685468